CLINICAL TRIAL: NCT00587262
Title: Scalar Localization of Cochlear Implant Electrode Array in Hearing Preservation Patients Using 64 Slice CT
Brief Title: Scalar Localization Cochlear Electrode Array Using 64 Slice CT
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lane, Professor of Radiology, College of Medicine, Mayo Clinic
Other Study IDs: 06-004832
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2009-09

CONDITIONS: Hearing Loss
Keywords: Cochlear; Hearing; High frequency hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, High-Frequency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Two pediatric participants with high frequency hearing loss post cochlear implant with either long or short electrode array.
- 2: Eight participants with high frequency hearing loss post cochlear implant with either short or long electrode array.
- 3: Fifteen participants from the existing Cochlear Implant data base.

SUMMARY:
Insertion of electrode array in scala vestibuli, rather than the preferred location within scala tympani, leads to loss of native hearing in those patients with isolated high-frequency hearing loss undergoing cochlear implantation.

DETAILED DESCRIPTION:
We aim to determine the surgical placement in patients with high frequency who had long electrode array insertions because they did not meet audiometric criteria for short array devices.

From this basis we will be able to determine if suboptimal insertion (e.g., in the scala vestibuli) leads to loss of low-frequency hearing in these patients. We also will look at the possibilities of using this data in predicting outcomes, modifying implant design, and perfecting surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Cochlear Implant Database.
* Patient has short or long electrode cochlear implant for high frequency hearing loss.

Exclusion Criteria:

* Inability to provide consent.
* Patients with underlying otospongiosis, extensive labyrinthitis ossificans or cochlear dysplasia. (These patients would have been identified with pre-operative imaging prior to cochlear implantation).

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Either part of the existing Cochlear Implant data base, or those persons who have had a Cochlear implant with either short or long electrode array who have had a high frequency hear loss.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The aim of our study is to determine surgical placement of the short electrode of cochlear implants in patients with high frequency loss. | Two years

SECONDARY OUTCOMES:
Determine the surgical placement in patients with high frequency who had long electrode array insertions because they did not meet audiometric criteria for short array devices. | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: John (Jack) I. Lane, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Lane JI, Witte RJ, Driscoll CL, Shallop JK, Beatty CW, Primak AN. Scalar localization of the electrode array after cochlear implantation: clinical experience using 64-slice multidetector computed tomography. Otol Neurotol. 2007 Aug;28(5):658-62. doi: 10.1097/MAO.0b013e3180686e26. PMID 17558341